CLINICAL TRIAL: NCT04113837
Title: Human Intervention Study for Validating the Influence of Regular Consumption of Foods With Improved Nutrient Profile on Cardiovascular Risk Factors
Brief Title: Human Intervention Study for Validating Foods With Improved Nutrient Profile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, Christine Dawczynski,PhD, PhD, University of Jena
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H9_19
Record Dates: First submitted 2019-10-01; First posted 2019-10-03 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2019-09

CONDITIONS: Cardiovascular Risk Factor
Keywords: foods, nutrient profile, dietary fiber, omega 3 fatty acids

STUDY DESIGN:
Intervention Model Description: The controlled, randomized, double-blind crossover study consists of a 4-week investigation periods with a 11-week wash-out period in between. At the beginning, participants are randomly allocated into the verum or the control/placebo group. After the wash-out phase the interventions are crossed between the groups and the respective food range is consumed also for four weeks.
Who Masked: Participant, Care Provider
Masking Description: The foods are offered in neutral packaging and are provided regularly by the study team. All personal (participants, care provider) are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- verum (Experimental): The food range is comprised of:
  sausages (1100 g per week / exchange of saturated fatty acids by long-chain unsaturated omega-3 fatty acids from fish oil (Maris Oil ED0222N rich in docosahexaenoic acid (DHA)), partially exchange of fat by plant protein (sesame)), eggs (3 eggs per week / 2 µg vitamin D per egg), 100 g mushrooms per day (5 µg Vitamin D/d), one bread per week (5 µg Vitamin D/d), bread rolls (16 g dietary fibers/d), 100 ml ice cream per week (exchange of sugar by xylitol), 3x 70 g pasta per week (3 x 10 g dietary fibers per week)
  Interventions: Dietary Supplement: food range
- control (Active Comparator): In the placebo period, the participants receive commercially available foods (sausages (raw, boiled and cooked varieties), eggs, mushrooms, bread, bread rolls, ice cream and pasta) with traditional nutrient profile.
  Interventions: Dietary Supplement: food range

INTERVENTIONS:
Dietary Supplement: food range — The food range is comprised of:
  sausages (1100 g per week) eggs (3 eggs per week), 100 g mushrooms per day, one bread per week, bread rolls, 100 ml ice cream per week, 3x 70 g pasta per week

SUMMARY:
The proposed intervention study is designed to evaluate the physiological impact of the regular consumption of the developed foods with improved nutrient profile (verum) in comparison to commercial available foods (control) by a controlled, randomized, double-blind crossover study with patients with measurable cardiovascular risk factors (LDL cholesterol ≥ 120 mg/dl (≥ 3 mmol/l) / Triacylglycerides ≥ 135 mg/dl (≥ 1,5 mmol/l)).

DETAILED DESCRIPTION:
The proposed intervention study is designed to evaluate the physiological impact of regularly consumption of the food range with improved nutrient profile (verum) in comparison to commercially available foods (control/placebo).

The controlled, randomized, double-blind crossover study consists of 4-week investigation periods with a 11-week wash-out period in between. Patients (men, female, n = 54 + 6) with measurable cardiovascular risk (LDL cholesterol ≥ 120 mg/dl (≥ 3 mmol/l) / triacylglycerides ≥ 135 mg/dl (≥ 1,5 mmol/l)), are involved.

The product range includes sausages (raw, boiled and cooked varieties) and pasta fortified with dietary fibers, fish oil and plant protein, resulting in a reduction of fat and energy content. Eggs, bread, bread rolls, and mushrooms with higher vitamin D content complete the innovative product range. Additionally, participants receive ice cream where sugar is replaced by xylite.

In the control period, the participants receive commercially available foods (sausages (raw, boiled and cooked varieties), pasta, eggs, bread, bread rolls, and mushrooms, ice cream) with traditional nutrient profile.

The products will be offered in neutral packaging and are provided regularly by the study team. All personal (participants, physicians) are blinded.

At the beginning, participants are randomly allocated into the verum or the control/placebo group. After the wash-out phase the interventions will be crossed between the groups and the respective products are consumed also for four weeks. In the run-in phase of the study, all patients are invited to a medical examination to ensure the fulfillment of inclusion criteria.

At the beginning and at the end of each study period baseline parameters (BMI, waist-to-hip ratio, blood pressure, bioelectrical impedance measurement) are assessed, lifestyle questionnaires are filled, and venous blood samples are collected for the determination of cardiovascular risk markers.

Subjects document their normal nutritional habits over seven days in a food frequency protocol (FFP) before start and finish of each period. In addition, patients keep a diary for the documentation of nutrition, medication and adverse effects over both study periods.

ELIGIBILITY:
Inclusion Criteria:

* females and males
* BMI < 30 kg/m2
* subjects must be able and willing to give written informed consent, and to comply with study procedures
* Participants following a traditional Western diet composed of dairy products, sausage, meat, fast foods, chocolate and snacks, cereals, vegetables, and fruits (PAL: 1.6)
* Precondition: Stable eating habits of at least one years before enrolment
* subjects with moderate elevated LDL cholesterol (≥ 3 mmol/l) and triacylglyceride concentrations (≥ 1.5 mmol/l) in plasma, without lipid-lowering medication
* stable dose of antihypertensive medication for > 3 months before study and during the entire study period or without antihypertensive medication
* subjects must have adequate fluency in the German language to complete the questionnaires and understand the nutritional recommendations

Exclusion Criteria:

* subjects with any acute or chronic disease (CVD, tumor, infection, other), gastrointestinal diseases, diabetes mellitus (type I and II), chronic renal disease, diseases of the parathyroid, diseases necessitating regular phlebotomies other chronic diseases which could affect the results of the present study
* use of prescription medicine which could affect results of the study, including systemic glucocorticoids
* intake of lipid-lowering drugs, diabetes medication, hormone replacement therapy
* estimated glomerular filtration (eGFR) rate < 60 ml/min
* weight loss (≤ 3 kg) or weight gain (≥ 3 kg) during the last three months before study begin
* pregnancy or lactation
* transfusion of blood in the last three months before blood sample taking
* use of dietary supplements incl. multivitamins, fish oil capsules, minerals, and trace elements (three months before and during the entire study period)
* vegetarians, vegans, food allergies (e.g. milk, nuts etc.)
* dependency on alcohol or drugs
* elite athletes (>10 hours of strenuous physical activity per week)
* simultaneous participation in other clinical studies
* inability (physically or psychologically) to comply with the procedures required by the protocol

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
LDL cholesterol | change from baseline after 4 weeks
  cardiovascular risk factor

SECONDARY OUTCOMES:
blood lipids | change from baseline after 4 weeks
  total cholesterol, HDL cholesterol, triglycerides in mmol/l
anthropometric data | change from baseline after 4 weeks
  body mass index (kg/m2)
blood pressure | change from baseline after 4 weeks
  systolic blood pressure (mm Hg) diastolic blood pressure (mmHg)
lipoprotein a | change from baseline after 4 weeks
  lipoprotein a (mg/l)
high-sensitive c-reactive protein | change from baseline after 4 weeks
  high-sensitive c-reactive protein (mg/dl)
homocysteine | change from baseline after 4 weeks
  homocysteine (µmol/l)
apolipoproteins | change from baseline after 4 weeks
  apolipoproteins A1, B (g/l)
glucose (fasting) | change from baseline after 4 weeks
  glucose (fasting) (mmol/l)
insulin (fasting) | change from baseline after 4 weeks
  insulin (fasting) (mU/l)
hemoglobin A1c (fasting) | change from baseline after 4 weeks
  hemoglobin A1c (fasting) (%)
malodialdehyde modified LDL cholesterol | change from baseline after 4 weeks
  malodialdehyde modified LDL cholesterol (U/l)
fatty acid distribution in plasma lipids | change from baseline after 4 weeks
  fatty acid distribution in plasma lipids (%FAME)
aspartate transaminase (AST) | change from baseline after 4 weeks
  aspartate transaminase (AST)
alanine transaminase (ALT) | change from baseline after 4 weeks
  alanine transaminase (ALT)
gamma-glutamyltransferase | change from baseline after 4 weeks
  gamma-glutamyltransferase (gGT)
Lactate dehydrogenase | change from baseline after 4 weeks
  Lactate dehydrogenase (LDH)
cholinesterase | change from baseline after 4 weeks
  cholinesterase
kalium | change from baseline after 4 weeks
  kalium (mmol/l)
transferrin | change from baseline after 4 weeks
  transferrin (g/l)
ferritin | change from baseline after 4 weeks
  ferritin (µg/l)
bioelectrical impedance | change from baseline after 4 weeks
  body water, body fat, lean body mass, extracellular mass (ECM), body cell mass (BCM)
vitamin A | change from baseline after 4 weeks
  vitamin A (mmol/l)
vitamin D | change from baseline after 4 weeks
  vitamin A (nmol/l)
vitamin E | change from baseline after 4 weeks
  vitamin E (µmol/l)
vitamin B1 | change from baseline after 4 weeks
  vitamin B1 (nmol/l)
vitamin B6 | change from baseline after 4 weeks
  vitamin B6 (nmol/l)
vitamin B12 | change from baseline after 4 weeks
  vitamin B12 (pmol/l)
vitamin B12 status | change from baseline after 4 weeks
  holotranscobalamine (pmol/l)
creatinine | change from baseline after 4 weeks
  creatinine (mmol/24 h)
natrium | change from baseline after 4 weeks
  natrium (mmol/24 h)
magnesium | change from baseline after 4 weeks
  magnesium (mmol/24 h)
zinc | change from baseline after 4 weeks
  zinc (µmol/24 h)
albumine | change from baseline after 4 weeks
  albumine (mg/l) (24 h urine)
uric acid | change from baseline after 4 weeks
  uric acid (mg/dl) (24 h urine)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Dawczynski, PhD, Principal Investigator — University of Jena
Locations (1):
- Friedrich Schiller University, Jena, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: recruiting — https://www.nuco.uni-jena.de/Rekrutierung.html